CLINICAL TRIAL: NCT00004437
Title: Phase II Study of the Multichannel Auditory Brain Stem Implant for Deafness Following Surgery for Neurofibromatosis 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Cochlear (Industry)
Purpose: Treatment
Other Study IDs: 199/13400; CC-FDR001283
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-01

CONDITIONS: Neurofibromatosis 2
Keywords: acoustic neuroma; genetic diseases and dysmorphic syndromes; hearing loss; neurofibromatosis; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic; Genetic Diseases, Inborn; Hearing Loss; Neurofibromatoses; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Device: Multichannel Auditory Brain Stem Implant

SUMMARY:
OBJECTIVES: I. Define the tonotopocity of multichannel brain stem stimulation and use this information to better program the auditory brain stem implant for an individual.

II. Optimize device fitting by combining monopolar and bipolar stimulation, and individual psychoacoustic channels for each patient, to increase the number of usable information channels for each patient and reduce or eliminate undesirable side effects.

III. Evaluate performance and learning effects using optimized fitting procedures.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients undergo surgery to remove the first side or second side tumor, during which the multichannel auditory brain stem implant is implanted. Initial stimulation is conducted 4-6 weeks after surgery.

Patients are followed every 3 months for the first year, then annually thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Confirmed diagnosis of neurofibromatosis type 2 Scheduled to undergo first side or second side tumor removal First side implantation performed only on patients with onset of symptoms prior to age 40 --Prior/Concurrent Therapy-- If a nonfunctional auditory brain stem implant (ABI) is present (implanted during the removal of a first side tumor), a multichannel ABI may be implanted during the removal of a second side tumor --Patient Characteristics-- English is the primary language

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Staller, Study Chair — Cochlear